CLINICAL TRIAL: NCT03176537
Title: Clinical, Microbiologic and Immunologic Profile of the Periodontal Condition in Hypogonadic Men
Brief Title: Periodontal Profile of Hypogonadic Men
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No eligible participants for the RCT were found
Sponsor: Universidade Federal do Paraná (Other)
Collaborators: Universidade Estadual Paulista - UNESP (Unknown); Universidade de Guarulhos (Unknown)
Responsible Party: Principal Investigator, Joao Paulo Steffens, PhD, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.906.729
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Periodontitis; Hypogonadism, Male
MeSH Terms: conditions — Periodontitis; Eunuchism

STUDY DESIGN:
Intervention Model Description: "Placebo" and "TRT" groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Gel, daily
  Interventions: Drug: Placebos
- TRT (Experimental): Testosterone Replacement Therapy
  Interventions: Drug: Testosterone gel

INTERVENTIONS:
Drug: Testosterone gel — Androgel (50mg testosterone), gel, daily
  Other Names: TRT
  Arms: TRT
Drug: Placebos — Placebo, gel, daily
  Arms: Placebo

SUMMARY:
The aim of this study is to assess if hypogonadic men with periodontitis benefit from testosterone replacement therapy before being submitted to periodontal treatment. Fifty hypogonadic men (Total Testosterone <200ng/dL) will be recruited from the Clinics Hospital at Federal University of Paraná and subjected to periodontal evaluation by a trained and calibrated researcher. The subjects presenting with periodontitis (assessed by clinical parameters) will be randomly allocated to "testosterone replacement therapy" (TRT) group or "placebo" for 3 months. After that time, all patients will receive nonsurgical periodontal treatment, which will be reassessed after 45 days. Clinical parameters (such as probing depth, gingival and plaque index, clinical attachment loss, bleeding on probing), sub gingival plaque and gingival crevicular fluid will be collected at baseline, just before therapy and 45 days after therapy.

ELIGIBILITY:
Inclusion Criteria: total testosterone <200ng/dL in two assessments; at least 20 teeth present.

-

Exclusion Criteria: systemic diseases such as hormonal, inflammatory and immune alterations.

-

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
CAL | 4.5 months
  Clinical Attachment Loss

SECONDARY OUTCOMES:
PPD | 4.5months
  probing pocket depth
PPD | 3months
  probing pocket depth
BOP | 3months
  bleeding on probing
BOP | 4.5months
  bleeding on probing
Micro-organisms concentration | 4.5months
  DNA hybridization - checkerboard
Micro-organisms concentration | 3months
  DNA hybridization - checkerboard
Concentration of inflammatory markers in crevicular fluid | 3months
  Multiplex assay
Concentration of inflammatory markers in crevicular fluid | 4.5 months
  Multiplex assay

CONTACTS AND LOCATIONS:
Overall Officials: Joao P Steffens, PhD, Principal Investigator — UFPR
Locations (1):
- Clínica de Odontologia da Universidade Federal do Paraná, Curitiba, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steffens JP, Coimbra LS, Rossa C Jr, Kantarci A, Van Dyke TE, Spolidorio LC. Androgen receptors and experimental bone loss - an in vivo and in vitro study. Bone. 2015 Dec;81:683-690. doi: 10.1016/j.bone.2015.10.001. Epub 2015 Oct 9. PMID 26450018
- [Background] Steffens JP, Wang X, Starr JR, Spolidorio LC, Van Dyke TE, Kantarci A. Associations Between Sex Hormone Levels and Periodontitis in Men: Results From NHANES III. J Periodontol. 2015 Oct;86(10):1116-25. doi: 10.1902/jop.2015.140530. Epub 2015 Jun 11. PMID 26062840
- [Background] Daltaban O, Saygun I, Bolu E. Periodontal status in men with hypergonadotropic hypogonadism: effects of testosterone deficiency. J Periodontol. 2006 Jul;77(7):1179-83. doi: 10.1902/jop.2006.050286. PMID 16805680